CLINICAL TRIAL: NCT06428526
Title: Effects of Afferent-specific Peripheral Electrical Stimulation (asES) on Sensorimotor Control and Tremor
Brief Title: Impact of Sensory Electrical Stimulation on Sensation and Tremor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Jose Pons, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00217703
Record Dates: First submitted 2024-04-30; First posted 2024-05-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Essential Tremor; Healthy Individuals
Keywords: Essential Tremor; Proprioception; Fine motor control; Electrical nerve stimulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous asES (Experimental): Participants will be administered transcutaneous afferent-specific electrical stimulation in the upper limb using conductive pads targeting the median and radial nerves at the wrist
  Interventions: Device: Continuous stimulation strategy; Device: Closed-loop stimulation strategy
- Percutaneous asES (Experimental): Participants will be administered percutaneous afferent-specific electrical stimulation in the upper limb using intramuscular leads targeting the flexor and extensor muscles of the wrist
  Interventions: Device: Continuous stimulation strategy; Device: Closed-loop stimulation strategy

INTERVENTIONS:
Device: Continuous stimulation strategy — Participants will be administered stimulation with a constant frequency stimulation.
Device: Closed-loop stimulation strategy — Participants will be administered with an activity-dependent stimulation.

SUMMARY:
The purpose of this study is to understand the acute, short-term and long-term impact of transcutaneous and/or percutaneous electrical stimulation with afferent-specific electrical stimulation (asES) on proprioception and fine motor control in the upper extremity. For this purpose, the researchers will use transcutaneous and/or percutaneous asES, high-density electromyography (HD-EMG), arm kinematic measurements, and standardized clinical assessments. This study will be conducted in healthy able-bodied individuals and patients with essential tremor (ET).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of afferent-specific electrical stimulation (asES), delivered either transcutaneous or percutaneous electrodes, on proprioception and fine motor control. The researchers will study the effect of asES in force perception, joint position perception, and touch sensitivity as proxies for proprioception. The researchers will also study the effect of asES on fine motor control by investigating the change in neural drive to the muscles before and after asES using the motor unit spike trains extracted from HD-EMG recordings. Furthermore, the researchers will also study the difference in effects of transcutaneous versus percutaneous asES on proprioception, fine motor control, and tremor in ET through HD-EMG and standard clinical measurements such as TETRAS and Perdue pegboard test. These results will help the researchers understand the acute, short-term, and long-term effects of various methods of asES delivery (transcutaneous or percutaneous) and their impact on proprioception and fine motor control.

Aim 1: Investigate the acute, short-term, and long-term effects of transcutaneous asES on proprioception and fine motor control. The overall goal of this study is to provide insight into the effect of transcutaneous stimulation of la afferent pathways targeted to modulate spinal reflexes in patients with ET to reduce tremors, which consequently might cause disruption in proprioception leading to changes in performance of fine motor control. The researchers hypothesize that asES might disrupt proprioception causing decreased performance in fine motor control tasks in the acute (during stimulation), and short-term (e.g., immediately following stimulation to 30 minutes post) but the effects will diminish in the long-term (up to 24 hours post stimulation) time periods.

Aim 2: Investigate the acute, short-term, and long-term effects of percutaneous asES on proprioception and fine motor control. The goal of this aim is to evaluate the effects of percutaneous asES to modulate Ia afferents and spinal reflexes to result in tremor reduction in ET, which consequently might cause disruption in proprioception leading to changes in performance of fine motor control. The researchers hypothesize that percutaneous asES will disrupt proprioception and fine motor control, but will also result in tremor reduction in the acute, short-term and long-term periods.

ELIGIBILITY:
Inclusion Criteria for Healthy Participants:

* Age from 18 to 80 years, inclusive
* No history of a brain and/or skull lesion
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* No neurological disorders
* No tremor
* Able to understand and speak English

Exclusion Criteria for Healthy Participants:

* History of significant head trauma (i.e., extended loss of consciousness, neurological damage)
* Known structural brain lesion
* Prior neurosurgical procedures
* Tremors (as determined by study team)
* Co-existence of other neurological diseases
* Parkinsonism
* Medical (e.g., cardiological, renal, hepatic, oncological) or psychiatric disease that would interfere with study procedures
* Pathology that could cause abnormal movements of extremities (e.g., epilepsy, stroke, marked arthritis, etc.)
* Inability to perform study tasks or assessments (e.g., follow instructions to stay still during asES procedures) or unable/unwilling to complete study forms
* Non-prescribed drug use or recreational marijuana use
* History of current substance abuse (exception: current nicotine use is allowed)
* Pregnancy
* Prisoners

Inclusion Criteria for ET Patients:

* Age from 18 to 80 years, inclusive
* No prior history of skull lesions or craniotomy
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* Diagnosis of ET (Tremor Research investigation Group criteria) by a physician
* At least moderate-severe tremor (based on the TETRAS Tremor Rating Scale) in an upper limb with pure flexion-extension wrist tremor during posture
* Stable medication doses for at least 30 days prior to study enrollment and during entire study period
* Able to understand and speak English

Exclusion Criteria for ET Patients:

* History of significant head trauma (i.e., extended loss of consciousness, neurological damage)
* Known structural brain lesion
* Prior neurosurgical procedures
* Mixed or complex tremors (as determined by study team)
* Co-existence of other neurological diseases
* Parkinsonism
* Medical (e.g., cardiological, renal, hepatic, oncological) or psychiatric disease that would - interfere with study procedures
* Pathology that could cause abnormal movements of extremities (e.g., epilepsy, stroke, marked arthritis, etc.)
* Inability to perform the study tasks or assessments (e.g., follow instructions to stay still during asES procedures) or unable/unwilling to complete study forms
* Non-prescribed drug use or recreational marijuana use
* History of current substance abuse (exception: current nicotine use is allowed)
* Pregnancy
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Force perception via force matching tasks | Assessment will be performed before, immediately after, and 30 minutes following the administration of the intervention in a single visit
  Force perception will be measured by evaluating the participant's ability to match a target force.
Position perception via position matching tasks | Assessment will be performed before, immediately after, and 30 minutes following the administration of the intervention in a single visit
  Position perception will be measured by evaluating the participant's ability to match a target joint position.
Touch perception using Semmes Weinstein monofilament testing | Assessment will be performed before, immediately after, and 30 minutes following the administration of the intervention in a single visit
  Touch perception will be assessed through Semmes-Weinstein monofilament testing. Roshen scores will be computed based on the filaments that are perceived by the participant. The range of Roschen scores can be from 0 -5. Higher scores mean better touch perception.
Fine motor control as assessed by visuomotor tracking performance | Assessment will be performed before, immediately after, and 30 minutes after the administration of the intervention in a single visit
  Fine motor control at the wrist and hands will be measured by evaluating the performance of the participants in tracking various forms of trajectory by moving their wrist and hand in flexion-extension movements.

SECONDARY OUTCOMES:
Tremor assessment using TETRAS | Assessment will be performed before, immediately after, and 30 minutes after the administration of the intervention in a single visit
  The Essential Tremor Rating Assessment Scale (TETRAS) will be used to quantify tremor of the participants. The TETRAS scale ranges from 0 - 64. Higher scores mean worse tremor in the participant.
Tremor assessment using arm kinematics | Assessment will be performed before, immediately after, and 30 minutes after the administration of the intervention in a single visit
  Upper limb kinematics using inertial measurement units (IMUs) will be used to quantify tremor of the participants. IMUs will be placed on the hand, forearm, and upper arm of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Pons, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No